CLINICAL TRIAL: NCT05165459
Title: Open Label Single Arm Proof of Concept Trial to Evaluate the Efficacy and Safety of Cytori Celution System in Chronic Non-Healing Venous Leg Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SZTE-CCS-LUL-01
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-12

CONDITIONS: Venous Leg Ulcer; Autologous Adipose Stromal Vascular Fraction; Adipose-Derived Mesenchymal Stem Cells; Mesenchymal Stem Cells
Keywords: Cytori Celution System
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cytori Celution System in Chronic Non-Healing venous Leg Ulcers (Experimental): On the screening visit, the study physician will assign one eligible ulcer, as the target ulcer. Target ulcer will be treated and followed up during the whole study period. After liposuction investigational device will be applied on the target ulcer. After completion of Day1 visit all subjects enter the observation period and will come back to 3 on-site visits on day 7 day 14 and day 28
  Interventions: Device: Venous leg ulcer treatment with adipous SVF

INTERVENTIONS:
Device: Venous leg ulcer treatment with adipous SVF — The Celution® System isolates approximately maximum 30 million SVF cells per 100 mL of adipose tissue to be processed. Approximately 1-3 million cells per injection (total 8-30) will be administered locally, in the target ulcer.

SUMMARY:
To evaluate the efficacy and safety of Cytori Celution System in Hungarian patients with chronic non-healing venous leg ulcers.

DETAILED DESCRIPTION:
This motive trial can help to establish routine application of this internationally widely used device at University of Szeged. The primary outcome is the reduction rate of the wound size. The treatment response will be calculated from wound size before and after treatment. Any adverse events related to the study device will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Males or females age ≥ 18
3. At least one venous chronic leg ulcer with the following condition 3.1. Ulcer is present beyond 2 months 3.2. Conservative treatment not leading to improvement 3.3. Wound size between ≥5 and ≤100 cm2
4. Ability to safely undergo tissue harvest that is anticipated to yield >100mL of adipose tissue at a site that is free from infection and injury
5. Able and willing to work with the doctor, adhere to therapeutic prescriptions and appear on prescribed examinations
6. Normal or clinically not significant abnormal values based on investigator judgement on white blood cell count (WBC), C-reactive protein (CRP), Platelets, international normalized ratio (INR), partial thromboplastin time (APTT), haemoglobin (Hgb), Renal and Liver function
7. Females of childbearing potential must have a negative pregnancy test at the Screen Visit
8. Females of childbearing potential must agree to use a highly effective method of birth control during the study. A highly effective method of birth control is defined as one which has a proven low failure rate of less than 1%

Exclusion Criteria:

1. More than 20% change in surface area of target ulcer between screening and enrollment visit.
2. There is bone involvement in case of ulcer
3. Patient with a history of bleeding disorder
4. Therapy for anticoagulation
5. Patient receiving corticosteroids, immunosuppressive or cytotoxic agents, and all systemic agents that can affect wound repair
6. Patient with any treatment that might interfere with the assessment of the study treatment
7. Pregnant or likely to become pregnant or lactating women
8. Participation in any type of clinical investigation concurrently or in the last 6 months
9. Positive for HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) and syphilis (results within 1 month are acceptable)
10. Any concurrent disease or condition that, in the opinion of the investigator, would make the patient unsuitable for the participation in the study.
11. Active cancer during chemotherapy or radiotherapy, or recent cancer, if the remission had place less than 5 years before joining the study (except basal cell skin cancer)
12. Patient currently undergoing dialysis for renal insufficiency (serum creatinine ≥2 mg/dL)
13. In the opinion of treating physician, patient not expected to survive beyond 30 days
14. Subjects with psychiatric conditions that are anticipated to result in protocol noncompliance
15. Uncontrolled chronic disease
16. Patient with history of severe alcohol or drug abuse
17. Lack of patient's cooperation
18. Use with blood thinners within 8 weeks of enrollment
19. Systemic treatments with a possible effect on ulcers within 4 weeks prior to enrollment with the following exceptions:

    1. Ustekinumab (within 16 weeks prior to enrollment)
    2. Adalimumab, infliximab, alefacept (within 8 weeks prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction rate of the wound size | 28 days
  The treatment response will be calculated from wound size before and after treatment.

SECONDARY OUTCOMES:
Wound closure at Day 28 | 28 days
  Percentage of patients achieving 50% wound closure at Day 28
Improvement of Quality of Life (QoL) - EQ-5D-5L | 28 days
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Improvement Wound pain | 28 days
  Improvement Wound pain visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Balázs Bende, MD, Principal Investigator — Szeged University; Lajos Kemény, Prof. Dr., Principal Investigator — Szeged University
Locations (1):
- University of Szeged Department of Dermatology and Allergology, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominici M, Le Blanc K, Mueller I, Slaper-Cortenbach I, Marini F, Krause D, Deans R, Keating A, Prockop Dj, Horwitz E. Minimal criteria for defining multipotent mesenchymal stromal cells. The International Society for Cellular Therapy position statement. Cytotherapy. 2006;8(4):315-7. doi: 10.1080/14653240600855905. PMID 16923606
- [Background] Le Blanc K, Ringden O. Immunomodulation by mesenchymal stem cells and clinical experience. J Intern Med. 2007 Nov;262(5):509-25. doi: 10.1111/j.1365-2796.2007.01844.x. PMID 17949362
- [Background] Galipeau J, Krampera M, Barrett J, Dazzi F, Deans RJ, DeBruijn J, Dominici M, Fibbe WE, Gee AP, Gimble JM, Hematti P, Koh MB, LeBlanc K, Martin I, McNiece IK, Mendicino M, Oh S, Ortiz L, Phinney DG, Planat V, Shi Y, Stroncek DF, Viswanathan S, Weiss DJ, Sensebe L. International Society for Cellular Therapy perspective on immune functional assays for mesenchymal stromal cells as potency release criterion for advanced phase clinical trials. Cytotherapy. 2016 Feb;18(2):151-9. doi: 10.1016/j.jcyt.2015.11.008. Epub 2015 Dec 23. PMID 26724220
- [Background] Horwitz EM, Le Blanc K, Dominici M, Mueller I, Slaper-Cortenbach I, Marini FC, Deans RJ, Krause DS, Keating A; International Society for Cellular Therapy. Clarification of the nomenclature for MSC: The International Society for Cellular Therapy position statement. Cytotherapy. 2005;7(5):393-5. doi: 10.1080/14653240500319234. PMID 16236628
- [Background] Meng X, Sun B, Xue M, Xu P, Hu F, Xiao Z. Comparative analysis of microRNA expression in human mesenchymal stem cells from umbilical cord and cord blood. Genomics. 2016 Apr;107(4):124-31. doi: 10.1016/j.ygeno.2016.02.006. Epub 2016 Feb 26. PMID 26921857
- [Background] Volz AC, Huber B, Kluger PJ. Adipose-derived stem cell differentiation as a basic tool for vascularized adipose tissue engineering. Differentiation. 2016 Jul-Aug;92(1-2):52-64. doi: 10.1016/j.diff.2016.02.003. Epub 2016 Mar 11. PMID 26976717
- [Background] Zachar V, Rasmussen JG, Fink T. Isolation and growth of adipose tissue-derived stem cells. Methods Mol Biol. 2011;698:37-49. doi: 10.1007/978-1-60761-999-4_4. PMID 21431509
- [Background] Schwartz RE, Reyes M, Koodie L, Jiang Y, Blackstad M, Lund T, Lenvik T, Johnson S, Hu WS, Verfaillie CM. Multipotent adult progenitor cells from bone marrow differentiate into functional hepatocyte-like cells. J Clin Invest. 2002 May;109(10):1291-302. doi: 10.1172/JCI15182. PMID 12021244
- [Background] Tang Y, Yasuhara T, Hara K, Matsukawa N, Maki M, Yu G, Xu L, Hess DC, Borlongan CV. Transplantation of bone marrow-derived stem cells: a promising therapy for stroke. Cell Transplant. 2007;16(2):159-69. PMID 17474297
- [Background] Aoi T, Stacey G. Impact of National and International Stem Cell Banking Initiatives on progress in the field of cell therapy: IABS-JST Joint Workshop: Summary for Session 5. Biologicals. 2015 Sep;43(5):399-401. doi: 10.1016/j.biologicals.2015.07.007. Epub 2015 Aug 24. PMID 26315652
- See also: Mesenchymal Stem Cells and Mononuclear Cells From Cord Blood: Cotransplantation Provides a Better Effect in Treating Myocardial Infarction — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4807668/
- See also: Wharton's Jelly-Derived Mesenchymal Stem Cells: Phenotypic Characterization and Optimizing Their Therapeutic Potential for Clinical Applications — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3709752/